CLINICAL TRIAL: NCT03721172
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study of the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Mild to Moderate Plaque Psoriasis
Brief Title: Apremilast as a Direct Treatment for Mild-to-moderate Plaque Psoriasis Versus Placebo: an Analysis of Clinical Safety and Efficacy
Acronym: ADVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-022; U1111-1218-8372 (Registry Identifier: WHO)
Record Dates: First submitted 2018-10-09; First posted 2018-10-26 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis
Keywords: Phase 3; Double-Blind; Efficacy; Safety; Apremilast; Otezla; CC-10004; Plaque Psoriasis; Mild; Moderate; Scalp; Nail; Itch
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular; Pruritus | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo-controlled Phase: (Experimental): Participants received placebo as oral tablets twice daily (BID) for up to 16 weeks (Week 0 to Week 16).
  Interventions: Other: Placebo
- Placebo-controlled Phase: Apremilast 30 mg (Experimental): Participants received apremilast 30 mg as oral tablets BID for up to 16 weeks (Week 0 to Week 16).
  Interventions: Drug: Apremilast
- Extension Phase: Apremilast 30 mg (Experimental): Eligible participants who completed the placebocontrolled phase entered the extension phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (Week 16 to Week 32).
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast, oral, twice daily
  Arms: Extension Phase: Apremilast 30 mg; Placebo-controlled Phase: Apremilast 30 mg
Other: Placebo — Placebo, oral, twice daily
  Arms: Placebo-controlled Phase:

SUMMARY:
This is a Phase 3, multicenter, randomized, placebo-controlled, double-blind study designed to evaluate the efficacy and safety of apremilast (CC-10004) in subjects with mild to moderate plaque psoriasis.

Approximately 574 subjects with mild to moderate plaque psoriasis will be randomized 1:1 to receive either apremilast 30 mg BID or placebo for the first 16 weeks.

DETAILED DESCRIPTION:
The study will consist of four phases:

* Screening Phase - up to 35 days
* Double-blind Placebo-controlled Phase - Weeks 0 to 16

  - Subjects will be randomly assigned to either apremilast 30 mg tablets orally BID or placebo tablets (identical in appearance to apremilast 30 mg tablets) orally BID.
* Apremilast Extension Phase - Weeks 16 to 32

  - All subjects will be switched to (or continue with) apremilast 30 mg BID. All subjects will maintain this dosing through Week 32.
* Observational Follow-up Phase - 4 weeks - Four-week Post-Treatment Observational Follow-up Phase for all subjects who complete the study or discontinue the study early.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must be male or female, ≥18 years of age at the time of signing the informed consent form (ICF).
2. Subject must have a diagnosis of chronic plaque psoriasis for at least 6 months prior to signing the ICF.
3. Subject must have a diagnosis of mild to moderate plaque psoriasis at both Screening and Baseline.
4. Subject must be inadequately controlled with or intolerant of at least one topical therapy at both Screening and Baseline.
5. Subject must be in good health (except for psoriasis) as judged by the investigator, based on medical history, physical examination, clinical laboratories, and urinalysis.
6. Subject must meet laboratory criteria.
7. Subject has not had prior exposure to biologics for the treatment of psoriatic arthritis or psoriasis, or any other condition that could impact the assessment of psoriasis.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subjects has any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.

2. Subject has hepatitis B surface antigen positive at Screening. 3. Subject has active tuberculosis (TB) or a history of incompletely treated TB.

4. Subject has history of positive human immunodeficiency virus (HIV), or has congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease).

5. Subject has hepatitis B surface antigen or anti-hepatitis C antibody positive at Screening.

6. Subject has prior history of suicide attempt at any time in the subject's life time or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent. 7. Subject has current or planned concurrent use of therapies that may have a possible effect on psoriasis during the course of the treatment phase of the trial.

8. Use of any investigational drug beginning 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).

9. Subject had prior treatment with apremilast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (64):
- United States (43):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - Northwest Arkansas Clinical Trials Center, PLLC / Hull Dermatology, Rogers, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - TCR Medical Corporation, San Diego, California
  - University of California San Francisco Psoriasis and Skin Treatment Center, San Francisco, California
  - Clinical Science Institute, Santa Monica, California
  - University of Colorado Hospital - Dermatology Clinic, Aurora, Colorado
  - Total Vein and Skin, LLC, Boynton Beach, Florida
  - Florida Academic Centers Research and Education, Coral Gables, Florida
  - International Dermatology Research, Miami, Florida
  - Center for Clinical and Cosmetic Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of South Florida - Carol and Frank Morsani Center for Advanced Health Care, Tampa, Florida
  - Atlanta Dermatology, Vein and Research Center, PC, Alpharetta, Georgia
  - Medical Dermatology Specialists, Inc. - Advanced Medical Research, Atlanta, Georgia
  - MedaPhase INC, Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Derm Associates, Rockville, Maryland
  - Lawrence Green, MD, LLC, Rockville, Maryland
  - ActivMed Practices & Research Inc, Beverly, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Central Dermatology, St Louis, Missouri
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Albert Einstein College of Medicine - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Temple University - Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah MidValley Dermatology, Murray, Utah
  - Virginia Clinical Research Inc, Norfolk, Virginia
  - Dermatology Center for Skin Health, Morgantown, West Virginia
- Canada (21):
  - Institute for Skin Advancement, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Chih-Ho Hong Medical, Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - SkinWise Dermatology, Winnipeg, Manitoba
  - Brunswick Dermatology Centre, Fredericton, New Brunswick
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research, Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Skin Center for Dermatology, Peterborough, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Sameh Hanna Medicine Professional Corporation DBA Dermatology on Bloor, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Dr Isabelle Delorme inc, Drummondville, Quebec
  - Dre Angelique Gagne-Henley M.D. Inc., Saint-Jérôme, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Stein Gold L, Papp K, Pariser D, Green L, Bhatia N, Sofen H, Albrecht L, Gooderham M, Chen M, Paris M, Wang Y, Callis Duffin K. Efficacy and safety of apremilast in patients with mild-to-moderate plaque psoriasis: Results of a phase 3, multicenter, randomized, double-blind, placebo-controlled trial. J Am Acad Dermatol. 2022 Jan;86(1):77-85. doi: 10.1016/j.jaad.2021.07.040. Epub 2021 Jul 31. PMID 34343599
- [Background] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 61 research centers in the United States and Canada from March 2019 to July 2020.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either apremilast or matched placebo for the first 16 weeks (placebo-controlled phase) of the study. At Week 16, eligible participants may have continued on active treatment by entering a 16 week extension phase (apremilast extension phase), total = 32 weeks.
Groups:
- Placebo-controlled Phase: Placebo: Participants received placebo as oral tablets twice daily (BID) for up to 16 weeks (Week 0 to Week 16).
- Extension Phase: Apremilast 30 mg: Eligible participants who completed the placebo-controlled phase entered the extension phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (Week 16 to Week 32).
Period: Placebo-controlled Phase
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Extension Phase: Apremilast 30 mg
Started | 298 | 297 | 0 (This arm was not included in the placebo-controlled phase.)
Received at Least 1 Dose of Treatment | 297 | 297 | 0 (This arm was not included in the placebo-controlled phase.)
Completed | 246 | 258 | 0 (This arm was not included in the placebo-controlled phase.)
Not Completed | 52 | 39 | 0
Not completed — Adverse Event | 7 | 7 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Lost to Follow-up | 15 | 13 | 0
Not completed — Withdrawal by Subject | 23 | 18 | 0
Not completed — Other | 3 | 0 | 0
Period: Apremilast Extension Phase
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Extension Phase: Apremilast 30 mg
Started | 0 (This arm was not included in the extension phase.) | 0 (This arm was not included in the extension phase.) | 503 (1 participant did not enter the extension phase due to physician decision.)
Received at Least 1 Dose | 0 (This arm was not included in the extension phase.) | 0 (This arm was not included in the extension phase.) | 503
Completed | 0 (This arm was not included in the extension phase.) | 0 (This arm was not included in the extension phase.) | 437
Not Completed | 0 | 0 | 66
Not completed — Adverse Event | 0 | 0 | 10
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 20
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 21
Not completed — Other | 0 | 0 | 3
Not completed — Other (Related to COVID-19) | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Total
Number analyzed (Participants) | 298 | 297 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (14.45) | 49.2 (14.65) | 48.7 (14.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 123 | 270
  Male | 151 | 174 | 325
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 31 | 64
  Not Hispanic or Latino | 260 | 264 | 524
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 7 | 8
  Asian | 18 | 15 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 17 | 14 | 31
  White | 257 | 254 | 511
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Static Physician Global Assessment (sPGA) Score [Count of Participants; unit: Participants] — The sPGA is a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 =severe. Scores incorporate an assessment by the Investigator of the severity of the 3 primary signs of the disease: erythema, scaling and plaque elevation.
  Participants
    2 (mild) | 91 | 91 | 182
    3 (moderate) | 207 | 206 | 413

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) Response at Week 16 During the Placebo-Controlled Phase
Description: The sPGA is a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 =severe. Scores incorporate an assessment by the Investigator of the severity of the 3 primary signs of the disease: erythema, scaling and plaque elevation.
  An sPGA response is defined as sPGA score of clear (0) or almost clear (1) and with at least a 2-point reduction from baseline at Week 16.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: Intent-to-treat (ITT) analysis set: all participants who were randomized into the placebo controlled phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 298 | 297
Percentage of participants | 4.1 [1.8 to 6.4] | 21.6 [16.7 to 26.4]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification were based on baseline sPGA (2 [mild] vs 3 [moderate]); Adjusted difference = 17.5, 95% CI 2-sided [12.2 to 22.8] — 2-sided 95% CIs based on the stratified Newcombe method. Stratification were based on baseline sPGA (2 [mild] vs 3 [moderate])

2. Secondary Outcome: Percentage of Participants With a ≥ 75 Percent (%) Improvement From Baseline in Affected Body Surface Area (BSA) at Week 16
Description: The BSA is a measurement of involved skin over the whole body. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand. The surface area of the whole body is made up of approximately 100 palms or "handprints" (each entire palmar surface or "handprint" equates to approximately 1% of total body surface area).
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set: all participants who were randomized in the placebo-controlled phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 298 | 297
Percentage of participants | 7.4 [4.2 to 10.6] | 33.0 [27.4 to 38.6]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification were based on baseline sPGA (2 [mild] vs 3 [moderate]); Adjusted difference = 25.6, 95% CI 2-sided [19.1 to 32.1] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Percentage of Affected BSA at Week 16
Description: The BSA is a measurement of involved skin over the whole body. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand. The surface area of the whole body is made up of approximately 100 palms or "handprints" (each entire palmar surface or "handprint" equates to approximately 1% of total body surface area).
  A negative change from baseline indicates a reduction of affected BSA.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set (all participants who were randomized) in the placebo-controlled phase with a baseline value and at least one post-baseline value at Week 16
Measure: Least Squares Mean (Standard Error); unit: Percentage change of affected BSA
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 249 | 261
Percentage change of affected BSA | -0.07 (0.24) | -3.45 (0.24)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Mixed-effect model for repeated measures; Least squares mean difference = -3.38, 95% CI 2-sided [-4.04 to -2.73], Standard Error of Mean 0.33

4. Secondary Outcome: Change From Baseline in Total Psoriasis Area Severity Index (PASI) Score at Week 16
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
  PASI scores range from 0 to 72, with higher scores reflecting greater disease severity.
  A negative change from baseline indicates an improvement of disease symptoms.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 249 | 261
Scores on a scale | -0.54 (0.20) | -3.47 (0.20)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Mixed-effect model for repeated measures; Least squares mean difference = -2.93, 95% CI 2-sided [-3.47 to -2.39], Standard Error of Mean 0.27

5. Secondary Outcome: Percentage of Participants Who Achieved BSA ≤ 3% for Participants With Baseline Affected BSA > 3% at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set (all participants who were randomized) in the placebo-controlled phase with baseline BSA > 3%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 255 | 245
Percentage of participants | 22.9 [17.4 to 28.4] | 61.0 [54.6 to 67.3]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification were based on baseline sPGA (2 [mild] vs 3 [moderate]); Adjusted difference = 38.0, 95% CI 2-sided [29.7 to 46.3] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants With ≥ 4-point Reduction From Baseline in Whole Body Itch Numeric Rating Scale (NRS) Score at Week 16 Who Had Baseline Whole Body Itch NRS ≥ 4
Description: The whole body itch NRS is a self-reported measure where participants were asked to assess whole body itch and select a number on a scale of 0-10, where 0 represents no itch, and 10 represents the worst imaginable itch. A reduction in score from baseline represents an improvement in symptoms.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set (all participants who were randomized) in the placebo-controlled phase with baseline whole body itch NRS score ≥ 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 249 | 253
Percentage of participants | 18.6 [13.4 to 23.7] | 43.2 [36.9 to 49.5]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification were based on baseline sPGA (2 [mild] vs 3 [moderate]); Adjusted difference = 24.7, 95% CI 2-sided [16.5 to 32.8] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants With a Scalp Physician Global Assessment (ScPGA) Response at Week 16 Among Participants With Baseline scPGA Score ≥ 2 at Week 16
Description: The ScPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an Investigator's assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation of the overall scalp.
  An ScPGA response is defined as and ScPGA score clear (0) or almost clear (1) with at least a 2-point reduction from baseline among participants with a baseline ScPGA score ≥ 2.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set (all participants who were randomized) in the placebo-controlled phase with baseline ScPGA Score ≥ 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 199 | 212
Percentage of participants | 16.6 [11.1 to 22.2] | 44.0 [37.1 to 51.0]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification were based on baseline sPGA (2 [mild] vs 3 [moderate]); Adjusted difference = 27.4, 95% CI 2-sided [18.6 to 36.3] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: The DLQI is a 10 item questionnaire dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from 0 (not at all) to 3 (very much). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No), and if "No," then the subject is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being 0 (not at all), 1 (a little) and 2 (a lot).
  Total scores have a possible range of 0 to 30, with 30 corresponding to the worst health-related quality of life, and 0 corresponding to the best score.
  A negative change from baseline indicates an improvement in health-related quality of life scores.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 249 | 261
Scores on a scale | -2.4 (0.3) | -5.2 (0.3)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Mixed-effect model for repeated measures; Least squares mean difference = -2.9, 95% CI 2-sided [-3.7 to -2.1], Standard Error of Mean 0.4

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A TEAE is any AE that occurs following administration of study treatment.
  Frequency of TEAEs was assessed as well as severity and treatment relatedness.
  A TEAE was considered severe based on the Investigator's assessment. A TEAE could be severe if it was serious or non-serious, had symptoms causing discomfort or pain, requiring medical or surgical attention or intervention, interfered with activities of daily life and if drug therapy was required.
Time Frame: Placebo: Day 1 to Week 16; Apremilast Day 1 to a maximum of Week 32 (plus 4 week safety follow-up)
Population: Safety analysis set: all randomized participants who received at least 1 dose of treatment. One participant randomized to the placebo group received apremilast and was therefore allocated to the apremilast group for the safety analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Apremalist: Placebo-controlled Phase and Extension Phase: All participants who received apremalist 30 mg as oral tablets BID in either the placebo-controlled phase (Week 0 to Week 16), the apremilast extension phase (Week 16 to Week 32), or both phases (Week 0 to Week 32)
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremalist: Placebo-controlled Phase and Extension Phase
Number analyzed (Participants) | 296 | 298 | 544
Participants
  Any TEAE | 139 | 195 | 351
  Severe TEAE | 2 | 8 | 24
  Treatment-related TEAE | 36 | 110 | 186

ADVERSE EVENTS:
Time Frame: Placebo: Day 1 to Week 16; Apremilast Day 1 to a maximum of Week 32 (plus 4 week safety follow-up)
Description: The safety analysis set includes all randomized participants who received at least 1 dose of investigational product. One participant randomized to the placebo group received apremilast and was therefore allocated to the apremilast group for the safety analysis.
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremalist: Placebo-controlled Phase and Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/296 | 0/298 | 0/544
Serious Adverse Events (participants affected / at risk) | 4/296 | 1/298 | 12/544
Other Adverse Events (participants affected / at risk) | 51/296 | 118/298 | 208/544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=296) | Placebo-controlled Phase: Apremilast 30 mg (N=298) | Apremalist: Placebo-controlled Phase and Extension Phase (N=544)
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 3
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Migraine without aura (Nervous system disorders) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=296) | Placebo-controlled Phase: Apremilast 30 mg (N=298) | Apremalist: Placebo-controlled Phase and Extension Phase (N=544)
Diarrhoea (Gastrointestinal disorders) | 15 | 49 | 78
Nausea (Gastrointestinal disorders) | 13 | 38 | 69
Nasopharyngitis (Infections and infestations) | 8 | 22 | 37
Upper respiratory tract infection (Infections and infestations) | 15 | 17 | 46
Headache (Nervous system disorders) | 15 | 39 | 70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03721172/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT03721172/SAP_001.pdf